CLINICAL TRIAL: NCT05899452
Title: Bubble Blowing As an Effective Method for Distraction During Pediatric IV Insertion: a Randomized Controlled Trial
Brief Title: Bubble Blowing As an Effective Distraction During Pediatric IV Insertion
Acronym: BubblesRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, James Chen, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H22-01928a
Record Dates: First submitted 2023-05-16; First posted 2023-06-12 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Pain; Anxiety
Keywords: Distraction; Bubbles; IV cannula insertion; Pediatric
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: One group will receive bubble distraction while another group will receive video distraction.
Masking Description: Cannot blind participants due to the nature of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bubbles (Experimental): Patient will receive bubble distraction method prior to and during the placement of their IV cannula
  Interventions: Behavioral: Bubble blowing (active)
- Video (Active Comparator): Patient will receive video distraction on an tablet computer prior to and during the placement of their IV cannula
  Interventions: Behavioral: Video distraction (passive)

INTERVENTIONS:
Behavioral: Bubble blowing (active) — Bubble blowing as a method of active distraction during painful procedure (insertion of an IV cannula)
  Arms: Bubbles
Behavioral: Video distraction (passive) — Video on a tablet computer as a method of passive distraction during painful procedure (insertion of an IV cannula)
  Arms: Video

SUMMARY:
Insertion of an IV cannula is a standard but potentially painful procedure. Distraction techniques are among the strategies used to alleviate this discomfort. The investigators are conducting a randomized controlled trial to assess whether bubble blowing is more effective than video distraction during IV insertions in young children in the medical imaging suite.

DETAILED DESCRIPTION:
Purpose:

To assess the effectiveness of two distraction techniques used to reduce the perceived pain of pediatric IV insertions, comparing bubble blowing versus watching videos.

Hypotheses:

1. Blowing bubbles will reduce perceived pain during IV insertions more than video watching in two- to five-year-olds.
2. Bubble-blowing will reduce child anxiety with IV insertion more than video watching.

Justification:

This study investigates whether bubble blowing is more effective in increasing patient comfort and reducing patient anxiety during IV insertions than the current standard practice. Managing patient comfort is essential because perioperative anxiety and pain lead to adverse outcomes, including prolonged induction of anesthesia, increased pain, increased incidence of postoperative delirium, and new onset negative behavioural changes.

Objectives:

* Primary Objective: To determine if bubble blowing reduces perceived pain during IV insertions more effectively than video watching in two- to five-year-old children.
* Secondary objectives: a) To compare child pain scores between bubble-blowing and video-watching groups; b) To quantify the rate of distress-free IV starts, as determined by the number of children with no worse than mildly uncomfortable.

Research Design:

This trial is designed as a randomized, controlled, superiority trial (RCT) involving children having an IV inserted in the medical imaging department; it aims to compare the effectiveness of distraction by bubble blowing versus video watching. Study participants will be randomized to either a bubble-blowing distraction group (Bubbles RCT intervention) or an iPad video-watching distraction group (Bubbles RCT control). A researcher not otherwise involved in the study will create a randomization schedule in blocks of four participants, and each participant's allocation will be concealed in envelopes. Participants and those conducting study procedures will be blinded to study allocation during recruitment. Next, the envelope will be opened, allocating the child to the control or experimental group to allow the pre-anesthetic consultation to explain what will happen and set family expectations.

Data collection procedures:

1. The research assistant (RA) will observe the child and their family and record a baseline modified Yale Preoperative Anxiety - Short Form (mYPAS-SF) score as soon as possible after consent is given.
2. Each participant will be randomized to bubble blowing group (Bubbles RCT intervention) or an iPad video-watching group (Bubbles RCT control). In both cases, the IV insertion will only occur after the topical anesthetic on the child's hands has had adequate time to take effect.
3. The Bubbles RCT control group will undergo the standard procedure for IV insertions in the medical imaging department but will utilize video distraction during IV insertions. Similarly, the Bubbles RCT intervention group will undergo the standard procedure for IV insertions in the medical imaging department but will utilize bubble-blowing distraction during IV insertion:

   1. The selected form of distraction (iPad video or Bubble blowing) will be active before the IV insertion procedure starts.
   2. The child will have their topical anesthetic removed and the IV placed quickly.
   3. The mYPAS-SF will be scored again by the RA observer as the patient enters the induction space or the clinician enters the patient's MRI anesthetic care unit (MRI-ACU) room. Pain will be assessed by the same observer using the Face Legs Activity Cry Consolability (FLACC) scale; this will be recorded twice during the IV insertion procedure (immediately before IV insertion and at the moment of skin penetration) and once more immediately after the IV insertion attempt is complete. The Bubbles RCT study ends at this point.
   4. If the IV insertion is unsuccessful on the first attempt, the provider will have discretion on how to proceed with the IV placement, including starting a second IV cannulation attempt after the final FLACC score is obtained or switching their induction of anesthesia modality.

Statistical Analysis: Participant demographics and characteristics will be tabulated and reported in a de-identified manner to protect participant privacy using descriptive statistics. Differences in FLACC pain scores between the two groups will be determined via a Wilcoxon rank sum test, as the investigators do not expect the data to be normally distributed. A linear regression model, controlling for age, sex, and baseline FLACC score, will be used to evaluate the superiority of the bubble-blowing technique. Similar analyses will be conducted for the mYPAS-SF scores.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of two to five years (i.e. ≥ two years to < six years) requiring an IV in the medical imaging department.

Exclusion Criteria:

* Children with existing vascular access (do not have an IV placed)
* Families who chose not to have topical anesthetic placed on their child's hands (will have a different amount of pain with the procedure than children who have had topical anesthetic)
* Children receiving anxiolytic premedication (will have reduced anxiety associated with the procedure)
* Children planned to undergo mask induction of anesthesia before IV placement (will not be awake to experience distraction method during IV insertion procedure)
* Children who had inadequate time for the local anesthetic cream/gel to take effect (pain will be experienced differently, and the effect of the local anesthetic will be more variable)

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Pain before IV insertion | at removal of topical anesthetic
  Observed pain score before IV insertion at timepoint 1 (removal of topical anesthetic), assessed using Face, Legs, Activity, Cry, Consolability (FLACC) scale (observer pain rating assessed on 5 dimensions with total scores ranging from 0 indicating no pain to 10 indicating highest pain).
Pain during IV insertion | at the moment of skin penetration
  Observed pain score during IV insertion at timepoint 2 (the moment of skin penetration) as measured by FLACC scale
Pain after IV insertion | once the IV insertion procedure is complete
  Observed pain score after IV insertion at timepoint 3 (once the IV insertion procedure is complete) as measured by FLACC scale

SECONDARY OUTCOMES:
Anxiety after consent | up to 5 minutes in waiting room immediately after consent
  Observed anxiety in waiting room as assessed using modified Yale Preoperative Anxiety Scale - Short Form (mYPAS-SF, observer anxiety rating, assessed on 4 dimensions with total scores ranging from 22.9 indicating minimal anxiety, to 100 indicating maximal anxiety)
Anxiety before IV insertion | between entering procedure room (or clinician approaching) until first IV insertion attempt
  Observed anxiety immediately before IV insertion procedure as assessed using mYPAS-SF

CONTACTS AND LOCATIONS:
Overall Officials: James Chen, MD, Principal Investigator — Provincial Health Services Authority British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Results will be presented at scientific conferences and published in peer-reviewed anesthesia journals. Once data collection is complete, a de-identified version of the data may be made available to other researchers. This is stated explicitly in the consent form, and participants are notified during the consent process that their de-identified data may be released to others for research purposes.
Supporting Information: Study Protocol, ICF
Time Frame: Once data collection is complete, de-identified data will be deposited in the University of British Columbia (UBC)'s Dataverse Repository. The study teams will keep research data for five years post-publication, as outlined in the UBC study data retention guidelines, after which it will be destroyed.
Access Criteria: Details have yet to be determined.

REFERENCES:
- [Background] Agbayani CG, Fortier MA, Kain ZN. Non-pharmacological methods of reducing perioperative anxiety in children. BJA Educ. 2020 Dec;20(12):424-430. doi: 10.1016/j.bjae.2020.08.003. Epub 2020 Oct 21. No abstract available. PMID 33456927
- [Background] Longobardi C, Prino LE, Fabris MA, Settanni M. Soap bubbles as a distraction technique in the management of pain, anxiety, and fear in children at the paediatric emergency room: A pilot study. Child Care Health Dev. 2019 Mar;45(2):300-305. doi: 10.1111/cch.12633. Epub 2018 Dec 12. PMID 30466144
- [Background] Chieng YJ, Chan WC, Klainin-Yobas P, He HG. Perioperative anxiety and postoperative pain in children and adolescents undergoing elective surgical procedures: a quantitative systematic review. J Adv Nurs. 2014 Feb;70(2):243-55. doi: 10.1111/jan.12205. Epub 2013 Jul 19. PMID 23865442
- [Background] Fortier MA, Del Rosario AM, Martin SR, Kain ZN. Perioperative anxiety in children. Paediatr Anaesth. 2010 Apr;20(4):318-22. doi: 10.1111/j.1460-9592.2010.03263.x. Epub 2010 Feb 23. PMID 20199609
- [Background] Vieco-Garcia A, Lopez-Picado A, Fuentes M, Francisco-Gonzalez L, Joyanes B, Soto C, Garcia de la Aldea A, Gonzalez-Perrino C, Aleo E. Comparison of different scales for the evaluation of anxiety and compliance with anesthetic induction in children undergoing scheduled major outpatient surgery. Perioper Med (Lond). 2021 Dec 14;10(1):58. doi: 10.1186/s13741-021-00228-x. PMID 34903293
- [Background] Jung MJ, Libaw JS, Ma K, Whitlock EL, Feiner JR, Sinskey JL. Pediatric Distraction on Induction of Anesthesia With Virtual Reality and Perioperative Anxiolysis: A Randomized Controlled Trial. Anesth Analg. 2021 Mar 1;132(3):798-806. doi: 10.1213/ANE.0000000000005004. PMID 32618627
- [Background] Krauss BS, Calligaris L, Green SM, Barbi E. Current concepts in management of pain in children in the emergency department. Lancet. 2016 Jan 2;387(10013):83-92. doi: 10.1016/S0140-6736(14)61686-X. Epub 2015 Jun 18. PMID 26095580
- [Background] Al-Yateem N, Brenner M, Shorrab AA, Docherty C. Play distraction versus pharmacological treatment to reduce anxiety levels in children undergoing day surgery: a randomized controlled non-inferiority trial. Child Care Health Dev. 2016 Jul;42(4):572-81. doi: 10.1111/cch.12343. Epub 2016 Apr 14. PMID 27080806
- [Background] Bahrololoomi Z, Sadeghiyeh T, Rezaei M, Maghsoudi N. The Effect of Breathing Exercise Using Bubble Blower on Anxiety and Pain during Inferior Alveolar Nerve Block in Children Aged 7 to 10 Years: A Crossover Randomized Clinical Trial. Pain Res Manag. 2022 Jan 17;2022:7817267. doi: 10.1155/2022/7817267. eCollection 2022. PMID 35082960
- [Background] Sridhar S, Suprabha BS, Shenoy R, Shwetha KT, Rao A. Effect of a relaxation training exercise on behaviour, anxiety, and pain during buccal infiltration anaesthesia in children: Randomized clinical trial. Int J Paediatr Dent. 2019 Sep;29(5):596-602. doi: 10.1111/ipd.12497. Epub 2019 Apr 8. PMID 30887592
- [Background] Lilik Lestari MP, Wanda D, Hayati H. The Effectiveness of Distraction (Cartoon-Patterned Clothes and Bubble-Blowing) on Pain and Anxiety in Preschool Children during Venipuncture in the Emergency Department. Compr Child Adolesc Nurs. 2017;40(sup1):22-28. doi: 10.1080/24694193.2017.1386967. PMID 29166202
- [Background] Kucuk Alemdar D, Yaman Aktas Y. The Use of the Buzzy, Jet Lidokaine, Bubble-blowing and Aromatherapy for Reducing Pediatric Pain, Stress and Fear Associated with Phlebotomy. J Pediatr Nurs. 2019 Mar-Apr;45:e64-e72. doi: 10.1016/j.pedn.2019.01.010. Epub 2019 Jan 30. PMID 30711327
- [Background] Ugucu G, Akdeniz Uysal D, Guzel Polat O, Artuvan Z, Polat Kulcu D, Aksu D, Gulgun Altintas M, Cetin H, Orekici Temel G. Effects of cartoon watching and bubble-blowing during venipuncture on pain, fear, and anxiety in children aged 6-8 years: A randomized experimental study. J Pediatr Nurs. 2022 Jul-Aug;65:e107-e114. doi: 10.1016/j.pedn.2022.03.016. Epub 2022 Apr 8. PMID 35410736
- [Background] Bellieni CV, Cordelli DM, Raffaelli M, Ricci B, Morgese G, Buonocore G. Analgesic effect of watching TV during venipuncture. Arch Dis Child. 2006 Dec;91(12):1015-7. doi: 10.1136/adc.2006.097246. Epub 2006 Aug 18. PMID 16920758
- [Background] Bergomi P, Scudeller L, Pintaldi S, Dal Molin A. Efficacy of Non-pharmacological Methods of Pain Management in Children Undergoing Venipuncture in a Pediatric Outpatient Clinic: A Randomized Controlled Trial of Audiovisual Distraction and External Cold and Vibration. J Pediatr Nurs. 2018 Sep-Oct;42:e66-e72. doi: 10.1016/j.pedn.2018.04.011. Epub 2018 May 1. PMID 29728296
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Jenkins BN, Fortier MA, Kaplan SH, Mayes LC, Kain ZN. Development of a short version of the modified Yale Preoperative Anxiety Scale. Anesth Analg. 2014 Sep;119(3):643-650. doi: 10.1213/ANE.0000000000000350. PMID 25010821
- [Background] West N, Christopher N, Stratton K, Gorges M, Brown Z. Reducing preoperative anxiety with Child Life preparation prior to intravenous induction of anesthesia: A randomized controlled trial. Paediatr Anaesth. 2020 Feb;30(2):168-180. doi: 10.1111/pan.13802. Epub 2020 Jan 8. PMID 31869478
- [Derived] Postles M, West N, Moxham L, Ramji J, Palm J, Morrison C, Gorges M, Chen J. The Effectiveness of Bubble-Blowing as a Distraction Technique During Pediatric Intravenous Cannulation: A Randomized Controlled Trial. Paediatr Anaesth. 2025 Aug;35(8):635-642. doi: 10.1111/pan.15138. Epub 2025 Jun 9. PMID 40488535
- See also: Pediatric Anesthesia Research Team website — http://bcchr.ca/PART